CLINICAL TRIAL: NCT07301736
Title: A Phase II Multinational, Multicentre, Double-blind, Randomised, Active-controlled, 3-way Cross-over Study to Evaluate the Therapeutic Equivalence of CHF5993 pMDI 100/6/12.5 µg HFA-152a Versus CHF5993 pMDI 100/6/12.5 µg HFA-134a in Subjects With Mild to Moderate Asthma
Brief Title: Therapeutic Equivalence of CHF5993 pMDI 100/6/12.5 µg HFA-152a in Subjects With Mild to Moderate Asthma
Acronym: TRECONY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993AA9-01; 2025-521456-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — norflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Treatment: CHF5993 pMDI (Pressurised Metered Dose Inhaler) with HFA-152a (Experimental): BDP (Beclometasone Dipropionate)/FF (Formoterol Fumarate)/GB (Glycopyrronium Bromide) 100/6/12.5 µg
  Interventions: Drug: CHF5993 pMDI with HFA-152a
- Reference Treatment 1: CHF5993 pMDI with HFA-134a (Active Comparator): BDP/FF/GB 100/6/12.5 µg
  Interventions: Drug: CHF5993 pMDI with HFA-134a
- Reference Treatment 2: CHF718 pMDI with HFA-134a (Active Comparator): BDP 100 µg
  Interventions: Drug: CHF718 pMDI with HFA-134a

INTERVENTIONS:
Drug: CHF5993 pMDI with HFA-152a — two puffs BID (twice daily)
  Arms: Test Treatment: CHF5993 pMDI (Pressurised Metered Dose Inhaler) with HFA-152a
Drug: CHF5993 pMDI with HFA-134a — two puffs BID
  Arms: Reference Treatment 1: CHF5993 pMDI with HFA-134a
Drug: CHF718 pMDI with HFA-134a — two puffs BID
  Arms: Reference Treatment 2: CHF718 pMDI with HFA-134a

SUMMARY:
This study will compare an asthma inhaler that uses a new climate friendly alternative propellant to an asthma inhaler with an existing propellant. We want to make sure both versions of the inhaler work the same way for people with mild to moderate asthma.

DETAILED DESCRIPTION:
This global study aims to compare whether the investigational inhaler with the new HFA-152a propellant is as safe, effective and well tolerated in patients with asthma as the inhalers that use the existing HFA-134a propellant. HFA-152a is a propellant gas that is designed to have a lower global warming potential and to be more climate friendly. The study will be conducted in Europe, Latin America, Ukraine, South Africa and United Kingdom. It is planned to randomize 468 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (18 ≤ age ≤ 75 years) with a diagnosis of Asthma for at least 6 months prior to screening and with diagnosis before the age of 50 years;
* Non-smokers, ex-smokers;
* Body mass index: within the range of 18.0 to 35.0 kg/m2 inclusive;
* Stable asthma therapy: a stable maintenance treatment for at least 4 weeks prior to screening with:

  1. low or medium doses of ICS (Inhaled Corticosteroids) alone; or
  2. low or medium doses of ICS + LABA (Long-acting β2-agonist) (fixed or free combination).
* Controlled or partly controlled based on an Asthma Control Questionnaire - 7 Items (ACQ-7) score <1.5 at screening and at randomisation.
* Pre-BD (Bronchodilator) FEV1 >40% and <90% of the predicted normal value, after appropriate wash out from BDs, at the Screening Visit (V1).
* A demonstrated increase in either FEV1 or forced vital capacity of >12% and >200 mL from baseline within 30 minutes (min) after inhalation of 400 µg salbutamol (i.e. albuterol) pMDI at the Screening Visit (V1).

Exclusion Criteria:

* History of near fatal asthma or hospitalisation for asthma in intensive care unit, inpatient setting or emergency room access for asthma in the previous 6 months prior to screening, which in the judgement of the Investigator may place the subjects at undue risk;
* Recent asthma exacerbation requiring systemic corticosteroids (SCSs), or emergency room admission or hospitalisation within 3 months prior to screening and/or during the run-in period ;
* Non-persistent asthma: exercise-induced, seasonal asthma (as the only asthma-related diagnosis) not requiring daily asthma control medicine;
* Asthma subjects currently treated with any of the following :

  1. High dose ICS;
  2. Long-acting muscarinic antagonist (LAMA);
  3. Systemic, depot or slow-release corticosteroids within 12 weeks prior to screening;
  4. Any other asthma treatments (e.g. cromolyn sodium, nedocromil sodium, leukotriene modifiers) within 4 weeks prior to screening;
  5. Any biologic therapy (e.g. omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab, tezepelumab) within 6 months prior to screening;
* Respiratory disorders other than asthma
* Lung resection;
* Lower respiratory tract infection;
* Lung cancer and history of lung cancer;
* Subjects with active cancer or a history of cancer (other than lungs) ;
* Patients who have clinically significant cardiovascular condition;
* Run-in compliance: e-Diary completion <75% and run-in treatment compliance <75% at randomisation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve from time zero to 4 hours (AUC0-4h) on Day 1 | Day 1
Change from baseline in pre-dose FEV1 on Day 28 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Piotr KUNA, MD, Principal Investigator — Barlicki University Hospital Medical University of Lodz, Poland
Locations (1):
- Elpida Trials - Parloes Hub, Dagenham, United Kingdom

IPD SHARING:
Plan to Share IPD: No